CLINICAL TRIAL: NCT01584102
Title: Better Together Healthy Caswell County: Randomized Controlled Trial Targeting Obesity-related Behaviors
Brief Title: Randomized Controlled Trial Targeting Obesity-related Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: VTech-2012-1
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Obesity
Keywords: Randomized controlled trial; obesity; community-based participatory research; minority health; rural health; health promotion
MeSH Terms: conditions — Obesity | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Behavioral: group fitness + education
- Group 2 (Active Comparator)
  Interventions: Behavioral: group fitness classes only

INTERVENTIONS:
Behavioral: group fitness + education — 15 weeks biweekly group fitness + 15 weekly nutrition and physical activity education
  Other Names: Eat Smart, Move More, Weigh Less
  Arms: Group 1
Behavioral: group fitness classes only — 15 weeks biweekly group fitness
  Arms: Group 2

SUMMARY:
The intervention included biweekly access to group fitness classes, with (Group 1) or without (Group 2) weekly nutrition and physical activity education sessions. Outcome measures were assessed at baseline and immediately post intervention and included BMI, waist circumference, blood pressure, physical activity and dietary behaviors, and psychosocial variables.

DETAILED DESCRIPTION:
This 15-week randomized controlled pilot study consisted of two groups. All participants received access to two group fitness classes per week, which were offered free of charge at the Caswell County Parks and Recreation Building. Zumba classes were offered one night a week, and the other evening was a 'potluck night' designed to increase participants exposure to a variety of other fitness classes such as floor aerobics, kickboxing, line dancing, and African dancing. Participants in the intervention group (Group 1) were enrolled in Eat Smart, Move More, Weigh Less (ESMMWL) where they received on hour weekly education classes on healthy eating and physical activity. The ESMMWL curriculum is a 15-week weight-management program that is delivered by local educators. Published research data were used to identify strategies that would lead to weight loss and/or weight maintenance. The program uses the Theory of Planned Behavior, and as such informs, empowers, and motivates participants to live mindfully as they make choices about eating and physical activity. The program provides opportunities for participants to keep a journal of healthy eating and physical activity behaviors.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age,
* English-speaking,
* No self-reported contraindications to exercise
* Eligible participants where scheduled an enrollment appointment. At this appointment, participants with blood pressure over 180/110 were directed to obtain immediate medical attention and were only eligible to enroll upon written consent from their physician

Exclusion Criteria:

* <18 years of age
* Non-English-speaking
* Self-reported contraindications to exercise
* Blood pressure over 180/110 without medical clearance

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Weight | 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M Zoellner, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Tech, Blacksburg, Virginia, United States